CLINICAL TRIAL: NCT02664129
Title: Video Self-observation as a Therapeutic Tool for Improving the Insight of Patients With Schizophrenia Disorders
Brief Title: Video as a Tool to Improve Insight in Schizophrenia
Acronym: VideoInsight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9545
Record Dates: First submitted 2016-01-11; First posted 2016-01-26 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2020-12

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; awareness; insight; video; self-observation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group with video (Experimental): 30 patients will watch the video of them in acute decompensation phase
  Interventions: Other: Video self-observation
- Control group without video (Sham Comparator): 30 patients will not watch the video of them in acute decompensation phase, they pass a standard interview with psychometric scales
  Interventions: Other: Non Self video observation

INTERVENTIONS:
Other: Video self-observation — Patients will watch the video of them in acute decompensation phase then they will be asked about their emotions, their understanding and awareness of mental illness
  Other Names: Group 1
  Arms: Experimental group with video
Other: Non Self video observation — Patients will not watch the video of them in acute decompensation phase.
  Other Names: Group 2
  Arms: Control group without video

SUMMARY:
The deficit of awareness of pathology (or insight) is a common symptom in patients with schizophrenia and has a negative impact on the prognosis of the disease. Current treatments aren't effective enough on this symptom (Pijnenbord et al., 2013).

Previous studies have shown a positive impact of videos of patients themselves on insight but they lacked power. This technique needs more investigation. The study aims to improve the patient's awareness of pathology with a video of themselves recorded in the acute phase of their illness. Patients will watch this video after clinical stabilization. This is a randomized controlled and single blinded trial. A population of 60 patients (30 in each group) will be included. The impact on the insight, symptomatology, treatment adherence and functional remission will be evaluated.

The video of patient is useful for a personalized clinical follow-up. Its use for therapeutic purposes would be innovative and could be extended to other applications in psychiatry, especially as this tool is readily available.

DETAILED DESCRIPTION:
In everyday practice in psychiatry, some interviews are filmed in order to follow the clinical course and for educational purposes. But the videos are not used as a therapeutic tool for patients. This research project focuses on the therapeutic potential of these videos and particularly on the awareness of patients of their disorder (insight). Patients hospitalized for decompensation of their schizophrenic pathology will be filmed during structured interviews. After clinical stabilization patients will be proposed to participate to this trial. A group of patients (G1) will watch the video recorded in the acute phase of their illness. A control group (G2) will have a usual care without video or specific therapy. 48 hours after, the clinical impact et the evolution of insight of patients will be evaluated. Then follow-up visits will also be provided at one and four months with the same clinical evaluation, plus an evaluation of treatment adherence and functional remission. This study also includes qualitative interviews for group 1 after watching the video to explore the experience of patients in this situation of self-confrontation. The autobiographical memory will also be studied in this protocol. Tolerance of this experience will be assessed by a monitoring of emotions, specifically depressive affects and suicidal ideation. Adverse events will be reported and patients will always have the access to a psychiatrist if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of schizophrenia or schizoaffective disorder according to the DSM 5
* Age between 18 and 65 years
* Patients initially hospitalized for acute decompensation of their schizophrenia or schizoaffective disorder according to the medical records and any medical certificates
* Patients who agreed to be filmed during a standardized interview at screening (in acute decompensation phase of the disease at the beginning of hospitalization)
* Clinical state compatible with the therapeutic experience and obtaining consent with a score on the scale of PANSS positive symptoms of less than 24

Exclusion Criteria:

* Mental impairment moderate to severe
* Central nervous system disease or severe head trauma
* Chronic alcohol dependence
* Patients hospitalized for a social problem or otherwise, without acute decompensation of their schizophrenia or schizoaffective disorder as assessed by the referring psychiatrist
* Patients deprived of liberty by judicial decision
* Pregnant and breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-12-08 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Unawareness of Mental Disorder (SUMD) | 48 hours
  Scale to assess Unawareness of Mental Disorder (SUMD)

SECONDARY OUTCOMES:
Insight | 48 hours
  Birchwood Insight Scale
Cognitif Insight | 48 hours
  Beck Cognitive Insight Scale
Positive Symptom | 48 hours
  Positive and Negative Symptom Scale
Negative Symptom | 48 hours
  Positive and Negative Symptom Scale
Depression | 48 hours
  Calgary Depression Scale for Schizophrenia
Autobiographical Memory | 48 hours
  Autobiographical Memory Test
Medication Adherence | 48 hours
  Medication Adherence Rating Scale
Functional Remission (FROGS scale) | 48 hours
  Evaluation of quality of daily life

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie SCHANDRIN, MD, Study Director — University hospital of Nîmes
Locations (2):
- France (2):
  - University Hospital of Montpellier, Montpellier
  - University Hospital of Nîmes, Nîmes

REFERENCES:
- [Derived] Schandrin A, Picot MC, Marin G, Andre M, Gardes J, Leger A, O'Donoghue B, Raffard S, Abbar M, Capdevielle D. Video self-confrontation as a therapeutic tool in schizophrenia: A randomized parallel-arm single-blind trial. Schizophr Res. 2022 Feb;240:103-112. doi: 10.1016/j.schres.2021.12.016. Epub 2022 Jan 3. PMID 34991040